CLINICAL TRIAL: NCT03599596
Title: Monthly Versus Two Doses of Ante-Natal Intermittent Preventive Treatment With Sulphadoxine-Pyrimethamine in University College Hospital
Brief Title: Monthly Versus Two Doses of Ante-Natal Intermittent Preventive Treatment With Sulphadoxine-Pyrimethamine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College Hospital, Ibadan (Other)
Responsible Party: Principal Investigator, Olaolu Olayinka ONI, Principal Investigator, University College Hospital, Ibadan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCHIbadan
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two doses of sulphadoxine-pyrimethamine (Active Comparator): 500mg of sulphadoxine and 25mg of pyrimethamine 3 tablets taken twice before delivery
  Interventions: Drug: Sulphadoxine-pyrimethamine
- Monthly doses of sulphadoxine-pyrimethamine (Active Comparator): 500mg of sulphadoxine and 25mg of pyrimethamine 3 tablets taken monthly delivery
  Interventions: Drug: Sulphadoxine-pyrimethamine

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine — Sulphadoxine-Pyrimethamine 500mg of Sulphadoxine and 25mg of Pyrimethamine 3tablets monthly until delivery
  Other Names: Vitadar
  Arms: Two doses of sulphadoxine-pyrimethamine
Drug: Sulphadoxine-pyrimethamine — Sulphadoxine-Pyrimethamine 500mg of Sulphadoxine and 25mg of Pyrimethamine 3tablets twice before delivery
  Other Names: Vitadar
  Arms: Monthly doses of sulphadoxine-pyrimethamine

SUMMARY:
Randomized controlled prospective comparative study

DETAILED DESCRIPTION:
This study is intended to be a randomized controlled comparative study conducted to compare the effect of monthly versus two doses of ante-natal intermittent preventive treatment with sulphadoxine-pyrimethamine

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Gestational age between 16 and 28weeks.
* No history of use of sulphadoxine-pyrimethamine prior to recruitment
* Not on any medication for prophylaxis

Exclusion Criteria:

* Anaemia
* HIV positive women
* Pre-existing medical conditions e.g diabetes mellitus, haemoglobinopathy, hypertension, kidney disease, heart disease, any endocrine disorder like hypo/hyperthyroidism, Cushing' disease, connective tissue disorders like systemic lupus erythematosus, antiphospholipid syndrome or any otherautoimmune disease with poor feto-maternal outcomes in pregnancy.
* History of Glucose -6-Phosphate Dehydrogenase (G6PD) deficiency in patient
* Allergy to sulphonamides or pyrimethamine.
* Non consenting patients
* Multiple gestations

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Sexes eligible for the study
Enrollment: 136 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Level of malaria parasitemia among pregnant women with monthly doses of sulphadoxine-pyrimethamine as compared to pregnant women with 2 doses of Intermittent Preventive Treatment of Malaria during Pregnancy with Sulphadoxine-Pyrimethamine (IPTp-SP). | 4 Months
  Number of participants with high level of malaria parasitemia in monthly doses of sulphadoxine-pyrimethamine group will be compared with the number of participants in 2 doses of IPTp-SP group.

SECONDARY OUTCOMES:
Prevalence of drug related adverse events associated with multiple doses of sulphadoxine pyrimethamine. | 4 Months
  Number of participants having drug related adverse events associated with multiple doses of sulphadoxine pyrimethamine will be noted.

REFERENCES:
- [Background] Agomo CO, Oyibo WA, Odukoya-Maije F. Parasitologic Assessment of Two-Dose and Monthly Intermittent Preventive Treatment of Malaria during Pregnancy with Sulphadoxine-Pyrimethamine (IPTP-SP) in Lagos, Nigeria. Malar Res Treat. 2011;2011:932895. doi: 10.4061/2011/932895. Epub 2011 Oct 26. PMID 22312575